CLINICAL TRIAL: NCT03033758
Title: Observational Study to Evaluate the Clinical Efficacy and Improved Quality of Life With the Administration of the Fixed Combination of Budesonide Formoterol, in Approximately 2000 Patients With Asthma
Brief Title: Evaluation of the Effectiveness and Quality of Life With the Administration of the Fixed Combination of Budesonide Formoterol in Greek Patients With Asthma During Routine Clinical Practice.
Acronym: BOREAS
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-HAL-EL-69
Record Dates: First submitted 2017-01-13; First posted 2017-01-27 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Asthma; Quality of Life
Keywords: comorbidities
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Budesonide/Formoterol treated patients — patients who are eligible to start their treatment with budesonide/formoterol therapy

SUMMARY:
This study will be conducted in Greek population. The patients who will be selected for study enrollment will receive inhaled combination of budesonide and formoterol fumarate dihydrate at doses 100 / 6mcg, 200 / 6mcg, 400/12 mcg through Elpenhlaler® device. The study end points will be efficacy and safety in patients with asthma.Additional study objectives will be quality of life, patient satisfaction, severe exacerbation and comorbidities.

DETAILED DESCRIPTION:
Asthma is a heterogeneous disease, usually characterized by chronic inflammation of the airways. Characterized by a history of respiratory symptoms such as wheezing, chest heaviness and cough symptoms that fluctuate over time, as well as variable airway obstruction.

Asthma is a common disease worldwide, the rates of which are increasing in children and adults. It is estimated that asthma affects 1-18% of the population in different countries. In Greece, which is a country with lower rates of asthma, it is estimated that 8.6% of the population suffers from the disease.

The diagnosis of asthma should be based on: Background with characteristic symptoms, signs variable airway obstruction, with tests for reversal of bronchial obstruction or other tests.

Long-term treatment of asthma has the following objectives 1. symptom control: achieve adequate control of symptoms and maintain normal activity levels 2. Risk Reduction: minimize risk of future exacerbations, permanent airflow obstruction and side effects from medication Pulmoton® is an inhaled combination of budesonide and formoterol fumarate dihydrate in portions 100 / 6mcg, 200 / 6mcg, 400/12 mcg, administered through Elpenhlaler® device, developed by ELPEN. It is approved as a bronchodilator in the treatment of asthma where administration of the combination (inhaled corticosteroid and long-beta2-agonist action) is appropriate in patients not adequately controlled with inhaled corticosteroids and 'as needed' inhaled beta2-agonists short-acting or patients already adequately controlled with both inhaled corticosteroids and long-acting beta2-agonists.

Pulmoton® not recommended for the initial treatment of asthma. The dosage of the individual components of Pulmoton® is separate and must be adjusted according to the severity of the condition. This should be considered not only at the beginning of therapy with fixed combination products, but also when adjusting the maintenance dosage.

The dose should be adjusted to the lowest possible, to achieve and maintain effective control of symptoms. Patients should be regularly reassessed by a doctor, so that the dose of Pulmoton® receiving remains optimal. When you achieve long-term control of symptoms with the lowest recommended dose, then the next step may be testing single administration of inhaled corticosteroid.

There are two alternatives for the treatment of asthma with Pulmoton®:

A. Pulmoton® maintenance therapy: Pulmoton® taken as regular maintenance treatment with a separate rapid-acting bronchodilator for relief of symptoms.

B. Pulmoton® maintenance and reliever therapy: Pulmoton® taken as regular maintenance and 'on demand' therapy to treat the symptoms.

A. Pulmoton® maintenance therapy:

Patients should be advised to always carry with them their fast-acting bronchodilator to use when there is a need for relief.

More information on the effectiveness and safety of the study drug, reported in the Summary of Product Characteristics (Summary of Product Characteristics (SmPC)

This prospective observational study aims to collect data regarding Pulmoton® from everyday clinical practice, improve the quality of life of patients and disease progression. The centers where the study will be approximately 100, both hospital and private pulmonary clinics will be held. Data will be collected for a period of 6 months from patients diagnosed with asthma not adequately controlled with inhaled corticosteroids and 'as needed' inhaled beta2-agonists short-acting or patients already adequately controlled on both inhaled corticosteroids and beta2-long-acting stimulants.

Data will be collected during the period of three (3) and six (6) months (± 2 weeks) from the initiation of treatment with inhaled combination include spirometry data, (FEV1, FVC, FEV / FVC), checklist ACQ, AQLQ questionnaire and questionnaire FSI 10, and details of any existing comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Patients about to start treatment with the inhaled combination of budesonide and formoterol fumarate dihydrate at doses 100 / 6mcg, 200 / 6mcg, 400/12 mcg, through Elpenhlaler device
* Regular treatment of asthma, wherein the administration of the combination (inhaled corticosteroid and long-action beta2-agonist) is appropriate
* Patients not adequately controlled with inhaled corticosteroids and 'as needed' inhaled beta2-agonists short-acting
* Patients who signed Informed Consent Patients eligible to follow the study procedures

Exclusion Criteria:

* Patients who will be treated out of SpC
* Patients without Informed Consent
* Patients not eligible to follow the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients about to start treatment with the inhaled combination of budesonide and formoterol fumarate dihydrate at doses 100 / 6mcg, 200 / 6mcg, 400/12 mcg, through Elpenhlaler device may be included in the study. Under current SPC, the Pulmoton indicated in the regular treatment of asthma, wherein the administration of the combination (inhaled corticosteroid and long-action beta2-agonist) is appropriate :
  * in patients not adequately controlled with inhaled corticosteroids and 'as needed' inhaled beta2-agonists short-acting
  * in patients already adequately controlled on both inhaled corticosteroids and long-acting beta2-agonists.
Sampling Method: Non-Probability Sample
Enrollment: 980 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
ACQ (change) | 6 months
  Evaluation of asthma control by varying the ACQ questionnaire from the start of treatment with Pulmoton® up over 6 months (± 2 weeks)

SECONDARY OUTCOMES:
FEV1 (change) | 6 months
  The change in FEV1
Quality of Life (change) | 6 months
  Evaluation of the quality of life of patients by changing the AQLQ questionnaire
FSI-10 (change) | 3 months
  Satisfaction of the patient to treatment with the inhaled combination budesonide formoterol through Elpenhlaler® device in either of the two dosages, after 3 months of treatment via FSI questionnaire 10
number of Adverse events | 6 months
  The incidence and frequency of exacerbations
Comorbidities | 6 months
  Recording of comorbidities which may exist and are known and the estimated change in the respective biochemical markers where they exist and are available)

CONTACTS AND LOCATIONS:
Locations (1):
- 7th Pulmonary Dept, Athens Chest Hospital, Athens, Mesogion Ave. 152, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: DOI: https://doi.org/10.18332/pne/144485 — https://doi.org/10.18332/pne/144485